CLINICAL TRIAL: NCT02926300
Title: Extension Study, An Open-labelled, Multi Center, Comparative Phase I/IIa Clinical Trials to Evaluate the Efficacy and Safety of FURESTEM-CD Inj. in Patients With Moderately Active Crohn's Disease
Brief Title: Long-term Safety and Efficacy of FURESTEM-CD Inj. in Patients With Moderately Active Crohn's Disease(CD)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kang Stem Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: KSTHD_FURESTEM-CD-EXT
Record Dates: First submitted 2015-11-11; First posted 2016-10-06 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2016-09

CONDITIONS: Crohn's Disease
Keywords: crohn's disease; stem cell therapy; inflammatory bowel disease; hUCB-MSC; UCB-MSC; Umbilical cord Blood; Rheumatoid Arthritis; RA; Stem cell; Cell therapy; Furestem; Mesenchymal stem cell; MSC
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: stem cells — IV infusion
  Other Names: FURESTEM-CD Inj.

SUMMARY:
The purpose of this clinical trial is to evaluate long-term safety and efficacy in patients who has history of FURESTEM-CD injection at least once.

DETAILED DESCRIPTION:
This study is an extended study of KSTHD_FURESTEM-CD phase 1 / 2a clinical trials in patients with moderate active Crohn's disease who had received at least once a FURESTEM-CD injection. The purpose of this clinical trial is to evaluate long-term safety and efficacy in patients for approximately 36 months (144 weeks).

ELIGIBILITY:
Inclusion Criteria:

* patients who has history of FURESTEM-CD Inj. injection at least once.
* patients who understand and voluntarily sign an informed consent form.

Exclusion Criteria:

* any other condition which the Principle Investigator judges would make subject unsuitable for study participation.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gender: Both Age Limits: 19years to 70years Healthy Volunteers?: No.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2015-11; Primary Completion 2021-10 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
all kinds of adverse events which occur during the clinical sutdy | 114 weeks
  Safety outcome

SECONDARY OUTCOMES:
ratio of patients who is applicable to CDAI<150 | 114 weeks
  Efficacy outcome
ratio of patients who reduce CDAI over 70 as contrasted witd baseline(V7) | 114 weeks
  Efficacy outcome

CONTACTS AND LOCATIONS:
Overall Officials: Suk-kyun Yang, Principal Investigator — Asan Medical Center
Locations (7):
- South Korea (7):
  - Inje University Haeundae Paik Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - Seoul National Universtiy Bundang Hospital, Seongnam-si
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Soeul National University Hospital, Soeul
  - The Catholic University of Korea, St. Vincent'S Hospital., Suwon